CLINICAL TRIAL: NCT03035409
Title: Effects of Anamorelin on Cancer-Related-Fatigue in Patients With Advanced Cancer
Brief Title: Anamorelin Hydrochloride, Physical Activity, and Nutritional Counseling in Decreasing Cancer-Related Fatigue in Patients With Incurable Metastatic or Recurrent Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0655; NCI-2017-00188 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0655 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignant Solid Neoplasm; C-Reactive Protein Measurement; Cancer Fatigue; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm; Weight Loss
MeSH Terms: conditions — Neoplasm Metastasis; Weight Loss | interventions — anamorelin; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive Care (anamorelin, physical activity, counseling) (Experimental): Patients receive anamorelin hydrochloride PO QD and undergo physical activity consisting of resistance exercises and a home walking program. Treatment continues for up to 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo nutritional counseling on day 21.
  Interventions: Drug: Anamorelin Hydrochloride; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Nutritional Assessment; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Anamorelin Hydrochloride — Given PO
  Other Names: RC-1291 HCl
Behavioral: Exercise Intervention — Undergo physical activity
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Nutritional Assessment — Undergo nutritional counseling
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well anamorelin hydrochloride, physical activity, and nutritional counseling work in decreasing cancer-related fatigue in patients with incurable solid tumors that have spread to other parts of the body or have come back. Anamorelin hydrochloride, physical activity, and nutritional counseling may help to decrease cancer-related fatigue in patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate changes in the Functional Assessment of Cancer Illness Therapy-Fatigue (FACIT-F) subscale score at day 43 +/- 3 days compared to baseline in patients with advanced cancer receiving oral anamorelin hydrochloride (anamorelin) 100 mg daily and standardized physical activity and nutritional counseling.

SECONDARY OBJECTIVES:

I. To examine the effects of anamorelin and standardized physical activity and nutritional counseling on health-related quality of life and patient reported outcomes as measured by the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF), Patient Reported Outcomes Measurement Information System (PROMIS) - Fatigue, Hospital Anxiety Depression Scale (HADS), Edmonton Symptom Assessment Scale (ESAS), Functional Assessment of Cancer Therapy (FACT-G) and its Functional Assessment of Anorexia/Cachexia Treatment (FAACT) subscale in these patients.

II. To examine the side effects and tolerability of anamorelin in these patients.

EXPLORATORY OBJECTIVES:

I. To explore the effects of anamorelin and standardized physical activity and nutritional counseling on muscle function (as measured by the 30 second chair stand test, 6 minute walk test, day time activity [accelerometer], body composition [as measured by INBODY], and resting energy expenditure [measured by indirect calorimetry]).

II. To characterize the effects of anamorelin on potential inflammatory biomarkers of cancer-related fatigue (CRF) (C-Reactive Protein [CRP], monocyte IL-6&R, TNF-a&R, IL-10, IL-8, IL-1&RA; IGF-1).

III. To explore the effects of anamorelin on sleep as measured by the Pittsburgh Sleep Quality Index (PSQI).

IV. To determine the association between change in FACIT-F scores and changes in muscle function, day time activity, and body composition, in patients with advanced cancer receiving oral anamorelin 100 mg daily and standardized physical activity and nutritional counseling.

OUTLINE:

Patients receive anamorelin hydrochloride orally (PO) once daily (QD) and undergo physical activity consisting of resistance exercises and a home walking program. Treatment continues for up to 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo nutritional counseling on day 21.

After completion of study treatment, patients are followed up on day 71.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of advanced cancer (metastatic or recurrent incurable solid tumors excluding prostate cancer)
* Presence of fatigue on FACIT-F subscale of =< 34 on a 0 to 52 scale (in which 52 = no fatigue and 0 = worst possible fatigue)
* Patient should describe fatigue as being present for a minimum of 2 weeks prior to screening
* CRP must be >= 3 mg/l in the absence of any other more likely cause of increased CRP like an infection or an autoimmune disorder
* No evidence of moderate to severe depression as determined by a HADS depression score of =< 13
* Presence of unintentional weight loss ranging from >= 2 - =< 15% in last 12 months
* Uncontrolled pain; if patient is on opioids for the treatment of cancer pain, he/she must have had no major dose change (> 25%) for at least 48 hours prior to study entry; the dose of morphine equivalent daily should not exceed 120 mg/day unless approved by the principal investigator (PI); change in opioid dose after study entry is allowed
* Patient must be willing to engage in telephone follow up with research staff
* Patient must have telephone access to be contacted by the research staff
* Hemoglobin level of >= 9 g/dL
* Estimated life expectancy of > 4 months at the time of screening
* Aspartate transaminase (AST) and alanine transaminase (ALT) levels =< 5 x upper limit of normal (ULN)

Exclusion Criteria:

* Major contraindications to anamorelin e.g. hypersensitivity
* Regularly engaged in moderate or vigorous-intensity exercise for at least 5 times a week
* Inability to complete the baseline assessment forms or to understand the recommendations for participation in the study
* Pregnant or lactating women, childbearing age women who are not on birth control; negative pregnancy test for women of childbearing potential, as defined by intact uterus and ovaries, and a history of menses within the last 12 months; pregnancy test to be performed no greater than 14 days prior to consent in study; in cases of women with elevated b-HCG, these candidates will be eligible to participate so long as the level of b-HCG is not consistent with pregnancy; women of childbearing potential need to be on or use contraception, or be abstinent during the study period; their male partners must also use contraception (condom) or maintain abstinence; birth controls specifications: women who are able to become pregnant must use birth control during the study and for 30 days after the last anamorelin dose; acceptable forms of birth control include barrier methods (such as condom or diaphragm) with spermicide
* Uncontrolled diabetes mellitus (fasting blood sugar > 200 mg/dl) at screening
* Male patients with a history of untreated hypogonadism
* Patients on drugs with strong CYP 3A4 inhibitors within the previous two weeks (ketoconazole, clarithromycin, itraconazole, nefazodone, telithromycin)
* Patients on drugs that may prolong the PR or QRS interval durations, such as any of the class I/sodium (Na+) channel blocking antiarrhythmic medications should be avoided (e.g. flecainide, procainamide, propafenone, quinidine)
* Patients with untreated clinically relevant hypothyroidism
* Patients currently on investigational therapies will be evaluated by the PI on a case by case basis and study participation approval will be obtained from the treating oncologist
* Patients with prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2026-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yennurajalingam S, Basen-Engquist K, Reuben JM, Fellman BM, Shete S, Maddi R, Williams JL, Dev R, Hui D, Bruera E. Anamorelin combined with physical activity, and nutritional counseling for cancer-related fatigue: a preliminary study. Support Care Cancer. 2022 Jan;30(1):497-509. doi: 10.1007/s00520-021-06463-8. Epub 2021 Jul 31. PMID 34331589
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with advanced cancer were recruited from the Supportive Care Center of MD Anderson Cancer Center with a fatigue score of < =34 on a 0 to 52 scale (FACIT-F) present for a minimum of 2 weeks before screening. Participants were recruited between February 2017 and December 2019.
Pre-assignment Details: 129 participants were enrolled in this study but 45 participants received the treatment. 84 participants did not receive treatment due to either screen failure or not eligible to receive treatment.
Groups:
- Anamorelin: Participants received Anamorelin 100mg tablet orally daily with standardized exercise prescription and nutritional support for 43 days.
Period: Overall Study
Arm/Group | Anamorelin
Started | 45
Day 15 | 28
Day 29 | 28
Day 43 | 28
Completed | 28
Not Completed | 17
Not completed — Adverse Event | 5
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Not completed — Non compliance | 4
Not completed — Patient was jittery | 1
Not completed — Did not like Questionnaire | 1
Not completed — Aspartate Aminotransferase increased | 1
Not completed — Did not like taking drugs | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anamorelin
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 64 [39 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28
Cancer Type [Count of Participants; unit: Participants]
  Lung | 17
  Gastrointestinal | 6
  Breast | 2
  Gynecological | 2
  Head and Neck | 1
Employment Status [Count of Participants; unit: Participants]
  Full time | 12
  Retired | 8
  Homemaker | 1
  Unemployed | 5
  Not Reported | 2
Marital Status [Count of Participants; unit: Participants]
  Divorced | 3
  Married | 21
  Single / never married | 2
  Widowed | 2

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
Description: FACIT Fatigue Subscale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The total score range is from 0-52. The higher the score, the lower the fatigue level. We calculated the mean change in FACIT-F fatigue subscale from baseline to Day 43.
Time Frame: Baseline up to day 43
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Anamorelin
Number analyzed (Participants) | 28
score on a scale | 4.89 [-0.18 to 9.96]

2. Secondary Outcome: The Edmonton Symptom Assessment Scale (ESAS)-Fatigue
Description: The Edmonton Symptom Assessment Scale (ESAS) is used to rate the intensity of ten common symptoms including fatigue experienced by cancer patients. The ESAS allows patients to rate the intensity of their fatigue using a 0-10 scale (0 = not at all, 10 = worst possible). The total ESAS score range from 0-100. The lower the score, the lower the fatigue level. We calculated the mean change in ESAS fatigue score from baseline to Day 43.
Time Frame: Baseline up to day 43
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Anamorelin
Number analyzed (Participants) | 28
score on a scale | -0.81 [-1.95 to 0.32]

3. Secondary Outcome: Multidimensional Fatigue Symptom Inventory-Short Form [MFSI-SF], General Fatigue
Description: The MFSI-SF is a 30-item multidimensional tool used to measure cancer related fatigue experienced in the past week. It consists of 5 empirically derived subscales: general, physical, emotional, mental and vigor. For each item, patients indicated their response on a 5-point Likert scale from 0 ("not at all") to 4 ("extremely fatigue"). Each of the 5 sub-scale score ranges from 0 to 24. The lower the score, the lower the fatigue level. We calculated the mean change in MFSI-SF general fatigue score from baseline to Day 43.
Time Frame: Baseline up to day 43
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Anamorelin
Number analyzed (Participants) | 28
score on a scale | -3.46 [-6.21 to -0.81]

4. Secondary Outcome: Multidimensional Fatigue Symptom Inventory-Short Form [MFSI-SF], Physical Fatigue
Description: The MFSI-SF is a 30-item multidimensional tool used to measure cancer related fatigue experienced in the past week. It consists of 5 empirically derived subscales: general, physical, emotional, mental and vigor. For each item, patients indicated their response on a 5-point Likert scale from 0 ("not at all") to 4 ("extremely fatigue"). Each of the 5 sub-scale score ranges from 0 to 24. The lower the score, the lower the fatigue level. We calculated the mean change in MFSI-SF physical fatigue score from baseline to Day 43.
Time Frame: Baseline up to day 43
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Anamorelin
Number analyzed (Participants) | 28
score on a scale | -0.39 [-2.34 to 1.56]

ADVERSE EVENTS:
Time Frame: adverse events were collected at baseline to Day 43
Arm/Group | Anamorelin
All-Cause Mortality (participants affected / at risk) | 2/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 10/28
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anamorelin (N=28)
Diarrhea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 10
Hyperglycemia (Endocrine disorders) | 5
Anorexia (Nervous system disorders) | 6
Insomnia (Nervous system disorders) | 6
Nausea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 3
Fever (General disorders) | 3
Pain (General disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3
Paresthesia (Skin and subcutaneous tissue disorders) | 3
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3
Arthalgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Rash maculopapular (Skin and subcutaneous tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Facial pain (Musculoskeletal and connective tissue disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Flatulence (Gastrointestinal disorders) | 2
Flushing (Nervous system disorders) | 2
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Hypertension (Vascular disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Hyponatremia (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT03035409/Prot_SAP_001.pdf